CLINICAL TRIAL: NCT01968330
Title: Postpartum Weight Loss in Obese Women Using a Sleep Intervention in a Group Prenatal Care Setting
Brief Title: Postpartum Weight Loss and Sleep Amongst Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Judette Louis, Assistant Professor College of Medicine Obstetrics and Gynecology Assistant Professor College of Public Health Community and Family Health, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00014850
Record Dates: First submitted 2013-10-18; First posted 2013-10-24 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Obesity; Sleep Disordered Breathing; Weight Loss; Postpartum; Insomnia
MeSH Terms: conditions — Obesity; Sleep Apnea Syndromes; Weight Loss; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Go!®to sleep (Experimental): Patients in the sleep intervention arm will undergo a sleep wellness program entitled Go!®to sleep as part of their group prenatal visits. This intervention is a six-week online program developed by the Cleveland clinic for non-pregnant patients suffering from insomnia. In collaboration with the Cleveland clinic sleep disorders center researchers will modify the program to fit the specific needs of a pregnant population. Subjects will receive access to the program and instructed on its use at their initial group prenatal visit. In subsequent visits subjects will be able to discuss their experience with the program.
  Interventions: Behavioral: Go!®to sleep
- Routine prenatal care (No Intervention): Patients in the routine prenatal care arm will complete prenatal care in a group setting and will not complete the sleep intervention.

INTERVENTIONS:
Behavioral: Go!®to sleep
  Arms: Go!®to sleep

SUMMARY:
This study will be a randomized controlled trial involving obese women obtaining prenatal care at an obstetric care clinic. Study subjects will undergo prenatal care in a group setting or prenatal care with a behavioral intervention to improve sleep. Anthropometric measurements, blood draws, questionnaires and at home sleep studies will be completed at three specified times (two antepartum and one postpartum). Primary outcome will be a comparison of postpartum weight loss amongst the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* • Pregnant female patients

  * Currently receiving obstetrical care at the TGH Health Park Genesis Clinic
  * Between in the second trimester at entry into the study
  * Overweight or obese defined as a pre-pregnancy body mass index greater than or equal to 25.0 kg/msquared
  * Over 18 years of age
  * Able to speak and understand as well as give informed consent in English
  * Have access to internet services
  * Have reported nightly sleep duration of <6.5 hours

Exclusion Criteria:

* • Under 18 years of age

  * Pre-existing type 1 or 2 diabetes mellitus
  * Pre-existing obstructive sleep apnea
  * Current use of sleep medication
  * Serious physical or mental illness or condition that would substantially interfere with participation in, or completion of, the entire intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Weight loss at 6 weeks postpartum. | six weeks postpartum
  The Primary objective of this study is to determine if a sleep intervention delivered in a group prenatal care setting of obese women can improve weight loss at one year postpartum (i.e. patient's ability to loose weight gained in pregnancy). This will be accomplished by:
  * Randomizing study subjects to groups with or without a sleep intervention component
  * Assessing weight, neck and abdominal circumference at each prenatal visit and at six weeks postpartum
  * Obtaining information regarding the patient's pre-pregnancy weight.
  * Assessing baseline sleep habits with at home polysomnography and actigraphy and repeating these measurements in the late third trimester as well as postpartum.
  * Assessing sleep habits through the Epworth Sleepiness scale and Pittsburgh Sleep Quality Index at baseline.
  * Obtaining qualitative feedback on the patient's experience with the sleep program and their sleep habits.

SECONDARY OUTCOMES:
Affects of improved sleep on insulin resistance and cholesterol levels | From the second trimester of pregnancy to six weeks postpartum
  The secondary objective will be to assess the affect of a sleep intervention on insulin resistance and cholesterol levels. This will be accomplished by:
  * Assessing glucose, insulin, HOMA, AUCgluc, leptin, adiponectin, total cholesterol, HDL, LDL, triglyceride levels at four time points in pregnancy and postpartum.
  * Completing the PRIME screen, a diet assessment tool, at approximately 20 weeks, 34 weeks and 6 and weeks postpartum
  * Assessing the neonates body composition at birth.

OTHER OUTCOMES:
Effect of improved sleep on mental health | Second trimester of pregnancy to six weeks postpartum.
  The tertiary objective will be to assess the affect of a sleep intervention on mental health This will be accomplished by
  * Perceived Stress Scale (PSS) at approximately 24 weeks, 38 weeks, and 6 weeks postpartum
  * Interpersonal Support Evaluation List (ISEL) at approximately 20 weeks gestation
  * Edinburgh Depression Scale at approximately 24 weeks and 6 weeks postpartum
  * COPE scale for ability to cope with stress at approximately 24 weeks, 38 weeks and 6 weeks postpartum
  * Obtaining qualitative feedback on the patient's mental health status throughout pregnancy.
Effect of sleep on breast milk composition | Second trimester of pregnancy to six weeks postpartum
  Breast milk will be collected from both arms at six weeks postpartum and evaluated for factors related to sleep including melatonin.

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Cain, MD, Study Chair — University of South Florida Department of OBGYN; Judette Louis, MD, MPH, Principal Investigator — University of South Florida Department of Obstetrics and Gynecology; Linda Odibo, Study Director — University of South Florida Department of Obstetrics and Gynecology
Locations (1):
- Tampa General Hospital Genesis Clinic, Tampa, Florida, United States

REFERENCES:
- [Derived] Cain MA, Brumley J, Louis-Jacques A, Drerup M, Stern M, Louis JM. A Pilot Study of a Sleep Intervention Delivered through Group Prenatal Care to Overweight and Obese Women. Behav Sleep Med. 2020 Jul-Aug;18(4):477-487. doi: 10.1080/15402002.2019.1613995. Epub 2019 May 25. PMID 31130005